CLINICAL TRIAL: NCT04830891
Title: A Volunteer Study to Collect Imaging Data for the Development and Validation of Intelligent Ultrasound ScanNav Anatomy PNB
Brief Title: A Volunteer Study to Collect Imaging Data for the Development and Validation of ScanNav Anatomy PNB
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2021_AG_05
Record Dates: First submitted 2021-03-24; First posted 2021-04-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Ultrasound Imaging of Anatomical Structures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-centre, prospective, non-randomised volunteer study to be undertaken in Intelligent Ultrasound's offices at Hodge House, 114-116 St Mary Street, Cardiff, CF10 1DY, UK.

DETAILED DESCRIPTION:
This is a single-centre, non-randomised, prospective study involving up to 100 participants. The data collected in this study will augment the data collected in ML2018_AG_01, ML2018_AG_02, IU2019_AG_03, and IU2020_AG_04.

Phase I Collect data from participants for each indicated block area. This set will be used to develop and verify models for the identification and highlighting of target anatomical structures on ultrasound images.

Phase II Validation will proceed by feeding the videos into the ScanNav AnatomyGuide system and recording the output anatomy highlighting, overlaid on the original ultrasound image. The overlaid video will be examined by experts to identify safety and performance issues.

ELIGIBILITY:
Inclusion Criteria:

Potential participants who meet the following criteria will be considered eligible for the study:

1. Male or female, at least 18 years of age;
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

Potential participants who meet the following criteria will NOT be eligible for the study:

1. Aged <18 years of age;
2. Unwilling or unable to provide informed consent;
3. Previous surgery or trauma to the affected area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be sourced initially from Intelligent Ultrasound's employees. If additional volunteers are required, adverts will be placed online. Intelligent Ultrasound will make cash payments of up to £40 to non-employee volunteers, to compensate them for their time
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Change in per-class Mean Intersection over Union (IoU) scores of deep-learning segmentation models compared to baseline models | 6 months
  The mean Intersection over Union will be computed for each class for each model trained with the enlarged dataset, using the existing unseen test data set. These scores will be compared with the scores from the existing baseline models to determine the effect of the enlarged training data

CONTACTS AND LOCATIONS:
Overall Officials: James Bowness, Principal Investigator — Clinical consultant, University of Oxford & Royal Gwent Hospital
Locations (1):
- Intelligent Ultrasound Limited, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No